CLINICAL TRIAL: NCT04310644
Title: Autonomic Neuropathy and Its Pathophysiology in Autoimmune Autonomic Neuropathies, Postural Orthostatic Tachycardia Syndrome and Ehlers Danlos Syndromes: Peripheral Autonomic Small Fiber Neuropathy or Central Autonomic Failure? Validation of the Malmö POTS Score and a Better Diagnosis of POTS in Patientes With Autnomic Failure (VaGeMAPS-3-step-Diag)
Brief Title: Autonomic Small Fiber Neuropathy and Ehlers Danlos Syndromes - Prospective Study and Registry
Acronym: ProANS
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Principal Investigator, Andrea Maier, Primary Investigator and attending physician, RWTH Aachen University
Other Study IDs: 19-016
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Autonomic Neuropathy; Ehlers-Danlos Syndrome Hypermobility Type; Small Fiber Neuropathy; Postural Tachycardia Syndrome
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Small Fiber Neuropathy; Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Postural Orthostatic Tachycardia Syndrome: Patients with orthostatic intolerance because of Postural orthostatic tachycardia syndrome diagnosed in our outpatient clinic by tilt table examination.
  Interventions: Other: No intervention planned, but all patients get our standart treatment
- Ehlers Danlos Syndrome: Patients with hypermobile or classical EDS who are already diagnosed including genetical testing for classical or vascular EDS and Marfan Syndromes
  Interventions: Other: No intervention planned, but all patients get our standart treatment
- Autoimmune autonomic neuropathy/Pure autonomic failure: Patients who have an autoimmune autonomic neuropathy based on clinical diagnosis and antibody testing in our outpatient clinic. Cardial MIBG Scintigraphy should have been performed.
  Interventions: Other: No intervention planned, but all patients get our standart treatment
- Healthy controls: Healthy controls with no documented cardiovascular or neurological disorders and no symtoms of autonomic failure/dizziness/fainting
- others: Patients who have comorbidities as mast cell activation syndrome, chronic fatigue and/or Post COVID syndrome, based on clinical diagnosis in our outpatient clinic.

INTERVENTIONS:
Other: No intervention planned, but all patients get our standart treatment — Patients are selected from clinical Routine and get our standart Treatment based on their disease
  Groups: Autoimmune autonomic neuropathy/Pure autonomic failure; Ehlers Danlos Syndrome; Postural Orthostatic Tachycardia Syndrome

SUMMARY:
We examine patients with different autonomic neuropathies and Ehlers Danlos syndromes compared to healthy controls at three different points over time (baseline, after 3 months and after 1.5 years) to gain knowledge about the course of this disease and understand its pathophysiology, with a focus on Small Fiber neuropathy. Moreover we will validate the german version of the Malmö POTS Score and establish an easy diagnostic scheme for patients in outpatient care.

DETAILED DESCRIPTION:
Inclusion of patients with autoimmune autonomic neuropathies/ pure autonomic failure, postural orthostatic tachycardia syndrome, small fiber neuropathies, Ehlers-Danlos syndromes, Mast cell activation syndrom, Chronic fatigue syndrome and PostCOVID syndrome in our Registry study with follow up visits. Comparison to healthy controls concerning selected examinations.

Planned examinations are laboratory tests, questionnaires on mental and physical health status and circulatory disorders, attention tests, tilt table testing, standing test, sweat function, investigation of small fiber function via quantitative sensory testing as well as the density of nerve fibers in the skin. Measurements are performed at baseline mostly in clinical routine and follow up visits are offered.

ELIGIBILITY:
Inclusion Criteria:

* autonomic neuropathy
* Postural orthostatic tachycardia syndrome
* hypermobile or classical Ehlers Danlos syndromes
* Chronic fatigue syndrome, mast cell activation syndrome and/or PostCOVID
* healty controls
* between 18-80 years
* in patients: diagnosis and clinical testing in our outpatient clinic
* German speaking

Exclusion Criteria:

* pregnancy
* Pacemaker or Deep brain Stimulation
* sensory or motor Polyneuropathy
* neurodegenerative disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will include patients with above mentioned disease who are diagnosed and treated in our outpatient clinic for autonomic disorders in Aachen, Germany.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | baseline, 3 months and 18 months
  Change in systolic and diastolic blood pressure over time
Heart frequency | baseline, 3 months and 18 months
  Change in heart frequency over time
Skin biopsy | baseline
  intraepithelial nerve fiber density between groups
Composite autonomic severity Score | baseline, 3 months and 18 months
  Change of the Score over time, the results are interpreted as normal (score=0), mild (score=1-3), moderate (score=4-6) or severe (score=7-10)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Maier, Principal Investigator — University Hospital, Aachen
Locations (1):
- University clinic RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Igharo D, Thiel JC, Rolke R, Akkaya M, Weis J, Katona I, Schulz JB, Maier A. Skin biopsy reveals generalized small fibre neuropathy in hypermobile Ehlers-Danlos syndromes. Eur J Neurol. 2023 Mar;30(3):719-728. doi: 10.1111/ene.15649. Epub 2022 Dec 13. PMID 36437696
- [Derived] Gerlach DA, Maier A, Manuel J, Bach A, Hoff A, Honemann JN, Heusser K, Voit D, Frahm J, Jordan J, Tank J. Real-Time Magnetic Resonance Imaging to Study Orthostatic Intolerance Mechanisms in Human Beings: Proof of Concept. J Am Heart Assoc. 2022 Nov;11(21):e026437. doi: 10.1161/JAHA.122.026437. Epub 2022 Oct 27. PMID 36300662
- See also: official homepage of our outpatient clinic for autonomic nervous system disorders — https://www.ukaachen.de/kliniken-institute/ans-ambulanz/die-ans-ambulanz.html
- See also: Paper Skin biopsy reveals generalized small fibre neuropathy in hypermobile Ehlers-Danlos syndromes — https://pubmed.ncbi.nlm.nih.gov/36437696/